CLINICAL TRIAL: NCT00870194
Title: A Comparison of Adding Exenatide With Switching to Exenatide in Patients With Type 2 Diabetes Experiencing Inadequate Glycemic Control With Sitagliptin Plus Metformin
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H8O-CR-GWDK
Record Dates: First submitted 2009-03-25; First posted 2009-03-27 (Estimated); Results first posted 2011-06-17 (Estimated); Last update posted 2015-04-09 (Estimated); Status verified 2015-03

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: diabetes; exenatide; Byetta; sitagliptin; Januvia; Amylin; Lilly
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Exenatide; Sitagliptin Phosphate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: exenatide and sitagliptin
- 2 (Placebo Comparator)
  Interventions: Drug: exenatide and placebo

INTERVENTIONS:
Drug: exenatide and sitagliptin — exenatide-subcutaneous injection, 5mcg (4 weeks) followed by 10mcg (16 weeks), twice a day; sitagliptin-100mg tablet orally once a day
  Other Names: exenatide-Byetta; sitagliptin-Januvia
  Arms: 1
Drug: exenatide and placebo — exenatide-subcutaneous injection, 5mcg (4 weeks) followed by 10mcg (16 weeks), twice a day; placebo-tablet orally once a day
  Other Names: exenatide-Byetta
  Arms: 2

SUMMARY:
The purpose of this study is to determine whether ceasing sitagliptin and switching to exenatide and metformin is non-inferior to adding exenatide to sitagliptin and metformin, in those patients with type 2 diabetes who are experiencing inadequate glycemic control with a combination of sitagliptin and metformin.

ELIGIBILITY:
Inclusion Criteria:

* Present with type 2 diabetes
* Patients have been treated with a stable dose of the following for at least 3 months prior to screening:

  * 100 mg/day sitagliptin and
  * ≥1500 mg/day metformin, or maximum tolerated dose (extended release or immediate-release).
* Have inadequate glycemic control as evidenced by an HbA1c between 7.1% and 9%, inclusive.
* Have a body mass index (BMI) ≥20 kg/m2 and <45 kg/m2

Exclusion Criteria:

* Are currently enrolled in, or discontinued within the last 30 days (or longer, if local guidelines require) from, a clinical trial involving an off-label use of an investigational drug or device, or concurrently enrolled in any other type of medical research judged not to be scientifically or medically compatible with this study.
* Have previously completed or withdrawn from this study or any other study investigating exenatide.
* Have a known allergy or hypersensitivity to exenatide, sitagliptin or excipients contained in exenatide or sitagliptin.
* Used drugs for weight loss (for example, orlistat, sibutramine, phenylpropanolamine, or similar over-the-counter medications) within 1 month of screening.
* Are currently treated with any of the following excluded medications:

  * Thiazolidinediones (TZD) within 3 months of screening.
  * Sulfonylurea (SU) within 3 months of screening.
  * Dipeptidyl peptidase-4 [DPP-4] inhibitors, with the exception of sitagliptin, within 3 months of screening.
  * Meglitinide derivatives (for example, repaglinide or nateglinide) within 3 months of screening.
  * Alpha-glucosidase inhibitors (for example, miglitol or acarbose) within 3 months of screening.
  * Exogenous insulin within the 3 months prior to screening.
  * Drugs that directly affect gastrointestinal motility, including, but not limited to: metoclopramide, cisapride, and chronic macrolide antibiotics.
  * Systemic corticosteroids (excluding topical and inhaled preparations) by oral, intravenous (IV), or intramuscular (IM) route used regularly (for longer than 1 month) or used within 1 month immediately prior to screening.
  * Any other oral antidiabetic (OAD) agent, other than sitagliptin or metformin, within 3 months prior to screening.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 255 (Actual)
Dates: Start 2009-03; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chief Medical Officer, MD, Study Director — Eli Lilly and Company
Locations (36):
- Argentina (2):
  - Research Site, Buenos Aires
  - Research Site, Morón
- Australia (3):
  - Research Site, Adelaide
  - Research Site, Geelong
  - Research Site, Melbourne
- Germany (15):
  - Research Site, Aschaffenburg
  - Research Site, Aßlar
  - Research Site, Beckum-Neubeckum
  - Research Site, Berlin
  - Research Site, Bosenheim
  - Research Site, Essen
  - Research Site, Falkensee
  - Research Site, Furth im Wald
  - Research Site, Grevenbroich
  - Research Site, Hohenmölsen
  - Research Site, Leipzig
  - Research Site, Neuwied
  - Research Site, Othmarschen
  - Research Site, Pohlheim
  - Research Site, Speyer
- Greece (2):
  - Research Site, Athens
  - Research Site, Thessaloniki
- India (5):
  - Research Site, Ahmedabad
  - Research Site, Bangalore
  - Research Site, Coimbatore
  - Research Site, Indore
  - Research Site, Jaipur
- Mexico (5):
  - Research Site, Coatzacoalcos
  - Research Site, Guadalajara
  - Research Site, Mérida
  - Research Site, Monterrey
  - Research Site, Tampico
- South Korea (4):
  - Research Site, Daegu
  - Research Site, Gwangju
  - Research Site, Seoul
  - Research Site, Ulsan

REFERENCES:
- [Derived] Violante R, Oliveira JH, Yoon KH, Reed VA, Yu MB, Bachmann OP, Ludemann J, Chan JY. A randomized non-inferiority study comparing the addition of exenatide twice daily to sitagliptin or switching from sitagliptin to exenatide twice daily in patients with type 2 diabetes experiencing inadequate glycaemic control on metformin and sitagliptin. Diabet Med. 2012 Nov;29(11):e417-24. doi: 10.1111/j.1464-5491.2012.03624.x. PMID 22375612

RESULTS

PARTICIPANT FLOW:
Groups:
- Exenatide + Placebo: Exenatide-subcutaneous injection, 5mcg (4 weeks) followed by 10mcg (16 weeks), twice a day; Placebo-tablet orally once a day.
- Exenatide + Sitagliptin: Exenatide-subcutaneous injection, 5mcg (4 weeks) followed by 10mcg (16 weeks), twice a day; Sitagliptin-100mg tablet orally once a day.
Period: Overall Study
Arm/Group | Exenatide + Placebo | Exenatide + Sitagliptin
Started | 127 | 128
Per Protocol Set | 97 | 111
Completed | 101 | 114
Not Completed | 26 | 14
Not completed — Adverse Event | 10 | 5
Not completed — Lack of Efficacy | 0 | 1
Not completed — Lost to Follow-up | 2 | 0
Not completed — Physician Decision | 3 | 1
Not completed — Protocol Violation | 3 | 3
Not completed — Entry Criteria Not Met | 1 | 2
Not completed — Subject Decision | 7 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Exenatide + Placebo | Exenatide + Sitagliptin | Total
Number analyzed (Participants) | 97 | 111 | 208
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 81 | 97 | 178
  >=65 years | 16 | 14 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.8 (10.97) | 54.6 (9.66) | 54.7 (10.27)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46 | 58 | 104
  Male | 51 | 53 | 104

OUTCOME MEASURES:

1. Primary Outcome: Change in HbA1c (Percent)
Description: Change in HbA1c from baseline to endpoint (Week 20); difference of base percent values [X% - Y%]
Time Frame: Baseline to 20 Weeks
Population: Per Protocol Set: the set of data generated by the subset of patients who sufficiently complied with the protocol to ensure that these data would be likely to exhibit the effects of treatment, according to the underlying scientific model.
Measure: Least Squares Mean (Standard Error); unit: Percent HbA1c
Arm/Group | Exenatide + Placebo | Exenatide + Sitagliptin
Number analyzed (Participants) | 97 | 111
Percent HbA1c | -0.38 (0.09) | -0.68 (0.08)
Statistical Analysis 1: Comparison: Exenatide + Placebo vs Exenatide + Sitagliptin; Test type: Non-Inferiority or Equivalence — Non-Inferiority Margin of 0.4%; p = .012, Mixed Model Repeated Measures
Statistical Analysis 2: Comparison: Exenatide + Placebo vs Exenatide + Sitagliptin; Power calculation: 80% assuming 200 patients (100 in each arm), no true difference and 1.0% standard deviation; Test type: Non-Inferiority or Equivalence — Non-inferiority margin of 0.4%; p = .012, Mixed Model Repeated Measures; Least Square Mean Difference = 0.30, 95% CI 2-sided [0.07 to 0.53], Standard Error of Mean 0.12 — Standard Error of the Least Square Mean

2. Secondary Outcome: Percentage of Patients Achieving HbA1c <=7.0%
Description: Percentage of patients whose baseline HbA1c was > 7.0% achieving HbA1c <=7.0% at endpoint (Week 20)
Time Frame: Baseline to 20 Weeks
Population: Patients in the Per Protocol Set whose baseline HbA1c was > 7.0%; Last Observation Carried Forward.Per Protocol Set: the set of data generated by the subset of patients who sufficiently complied with the protocol to ensure that these data would be likely to exhibit the effects of treatment, according to the underlying scientific model.
Measure: Number; unit: Percentage
Arm/Group | Exenatide + Placebo | Exenatide + Sitagliptin
Number analyzed (Participants) | 88 | 106
Percentage | 29.5 | 44.3
Statistical Analysis 1: Comparison: Exenatide + Placebo vs Exenatide + Sitagliptin; Test type: Superiority or Other; p = .038, Fisher's Exact Test

3. Secondary Outcome: Percentage of Patients Achieving HbA1c <7.0%
Description: Percentage of patients whose baseline HbA1c was >=7.0% achieving HbA1c <7.0% at endpoint (Week 20)
Time Frame: Baseline to 20 Weeks
Population: Patients in the Per Protocol Set whose baseline HbA1c was >= 7.0%; Last Observation Carried Forward. Per Protocol Set: the set of data generated by the subset of patients who sufficiently complied with the protocol to ensure that these data would be likely to exhibit the effects of treatment, according to the underlying scientific model.
Measure: Number; unit: Percentage
Arm/Group | Exenatide + Placebo | Exenatide + Sitagliptin
Number analyzed (Participants) | 94 | 108
Percentage | 26.6 | 41.7
Statistical Analysis 1: Comparison: Exenatide + Placebo vs Exenatide + Sitagliptin; Test type: Superiority or Other; p = .027, Fisher's Exact Test

4. Secondary Outcome: Percentage of Patients Achieving HbA1c <=6.5%
Description: Percentage of patients whose baseline HbA1c was > 6.5% achieving HbA1c <=6.5% at endpoint (Week 20)
Time Frame: Baseline to 20 Weeks
Population: Patients in the Per Protocol Set whose baseline HbA1c was > 6.5%; Last Observation Carried Forward. Per Protocol Set: the set of data generated by the subset of patients who sufficiently complied with the protocol to ensure that these data would be likely to exhibit the effects of treatment, according to the underlying scientific model.
Measure: Number; unit: Percentage
Arm/Group | Exenatide + Placebo | Exenatide + Sitagliptin
Number analyzed (Participants) | 97 | 111
Percentage | 16.5 | 20.7
Statistical Analysis 1: Comparison: Exenatide + Placebo vs Exenatide + Sitagliptin; Test type: Superiority or Other; p = .480, Fisher's Exact Test

5. Secondary Outcome: Change in FSG (mmol/L)
Description: Change in fasting serum glucose (FSG) from baseline to endpoint (Week 20)
Time Frame: Baseline to 20 Weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Exenatide + Placebo | Exenatide + Sitagliptin
Number analyzed (Participants) | 93 | 106
mmol/L | 0.06 (0.23) | -0.55 (0.21)
Statistical Analysis 1: Comparison: Exenatide + Placebo vs Exenatide + Sitagliptin; Test type: Superiority or Other; p = .038, ANCOVA

6. Secondary Outcome: Change in Body Weight (kg)
Description: Change in body weight from baseline to endpoint (Week 20)
Time Frame: Baseline to 20 Weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: kg
Arm/Group | Exenatide + Placebo | Exenatide + Sitagliptin
Number analyzed (Participants) | 97 | 111
kg | -2.58 (0.25) | -2.20 (0.24)
Statistical Analysis 1: Comparison: Exenatide + Placebo vs Exenatide + Sitagliptin; Test type: Superiority or Other; p = .266, Mixed Model Repeated Measures

7. Secondary Outcome: Change in Waist Circumference (cm)
Description: Change in waist circumference from baseline to endpoint (Week 20)
Time Frame: Baseline to 20 Weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: cm
Arm/Group | Exenatide + Placebo | Exenatide + Sitagliptin
Number analyzed (Participants) | 96 | 111
cm | -3.25 (0.40) | -2.36 (0.37)
Statistical Analysis 1: Comparison: Exenatide + Placebo vs Exenatide + Sitagliptin; Test type: Superiority or Other; p = .095, Mixed Model Repeated Measures

8. Secondary Outcome: Waist-to-Hip Ratio
Description: Change in waist-to-hip ratio from baseline to endpoint (Week20)
Time Frame: Baseline to 20 Weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Ratio
Arm/Group | Exenatide + Placebo | Exenatide + Sitagliptin
Number analyzed (Participants) | 96 | 111
Ratio | -0.01 (0.00) | -0.00 (0.00)
Statistical Analysis 1: Comparison: Exenatide + Placebo vs Exenatide + Sitagliptin; Test type: Superiority or Other; p = .567, Mixed Model Repeated Measures

9. Secondary Outcome: SMBG (mmol/L)
Description: 7 point Self Monitored Blood Glucose Profiles - daily mean value (Week 20)
Time Frame: Baseline to 20 Weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Exenatide + Placebo | Exenatide + Sitagliptin
Number analyzed (Participants) | 50 | 71
mmol/L | 8.57 (0.26) | 8.16 (0.22)
Statistical Analysis 1: Comparison: Exenatide + Placebo vs Exenatide + Sitagliptin; Test type: Superiority or Other; p = .207, Mixed Model Repeated Measures

10. Secondary Outcome: Change in Triglycerides (mmol/L)
Description: Change in triglycerides from baseline to endpoint (Week 20)
Time Frame: Baseline to 20 Weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Exenatide + Placebo | Exenatide + Sitagliptin
Number analyzed (Participants) | 96 | 109
mmol/L | 0.17 (0.10) | -0.07 (0.09)
Statistical Analysis 1: Comparison: Exenatide + Placebo vs Exenatide + Sitagliptin; Test type: Superiority or Other; p = .055, ANCOVA

11. Secondary Outcome: Change in HDL (mmol/L)
Description: Change in high-density lipoprotein (HDL) cholesterol from baseline to endpoint (Week 20)
Time Frame: Baseline to 20 Weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Exenatide + Placebo | Exenatide + Sitagliptin
Number analyzed (Participants) | 96 | 109
mmol/L | -0.03 (0.02) | -0.01 (0.02)
Statistical Analysis 1: Comparison: Exenatide + Placebo vs Exenatide + Sitagliptin; Test type: Superiority or Other; p = .269, ANCOVA

12. Secondary Outcome: Change in LDL (mmol/L)
Description: Change in low-density lipoprotein (LDL) cholesterol from baseline to endpoint (Week 20)
Time Frame: Baseline to 20 Weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Exenatide + Placebo | Exenatide + Sitagliptin
Number analyzed (Participants) | 90 | 98
mmol/L | 0.06 (0.06) | 0.10 (0.06)
Statistical Analysis 1: Comparison: Exenatide + Placebo vs Exenatide + Sitagliptin; Test type: Superiority or Other; p = .622, ANCOVA

13. Secondary Outcome: Change in Total Cholesterol (mmol/L)
Description: Change in total cholesterol from baseline to endpoint (Week 20)
Time Frame: Baseline to 20 Weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Exenatide + Placebo | Exenatide + Sitagliptin
Number analyzed (Participants) | 96 | 109
mmol/L | 0.09 (0.07) | 0.08 (0.07)
Statistical Analysis 1: Comparison: Exenatide + Placebo vs Exenatide + Sitagliptin; Test type: Superiority or Other; p = .888, ANCOVA

14. Secondary Outcome: Incidence of Hypoglycemia (Overall)
Description: Incidence of hypoglycemic episodes experienced overall during the study
Time Frame: Baseline to 20 Weeks
Population: As Treated Patients; Hypoglycemia defined as: patient experiencing a sign or symptom associated with hypoglycemia that is either self-treated or resolves on its own; not confirmed with blood glucose values.
Measure: Number; unit: Participants
Arm/Group | Exenatide + Placebo | Exenatide + Sitagliptin
Number analyzed (Participants) | 127 | 128
Participants | 5 | 10
Statistical Analysis 1: Comparison: Exenatide + Placebo vs Exenatide + Sitagliptin; Test type: Superiority or Other; p = .287, Fisher's Exact Test

15. Secondary Outcome: Incidence of Severe Hypoglycemia(Overall)
Description: Incidence of severe hypoglycemia experienced overall during the study
Time Frame: Baseline to 20 Weeks
Population: As Treated Patients; Severe hypo:symptoms consistent with hypoglycemia resulting in loss of consciousness or seizure with prompt recovery in response to administration of glucagon or glucose;or documented hypoglycemia (BG< 3.0 mmol/L [54/mg/dL]) requiring the assistance of another person because of severe impairment in consciousness or behavior
Measure: Number; unit: Participants
Arm/Group | Exenatide + Placebo | Exenatide + Sitagliptin
Number analyzed (Participants) | 127 | 128
Participants | 1 | 0
Statistical Analysis 1: Comparison: Exenatide + Placebo vs Exenatide + Sitagliptin; Test type: Superiority or Other; p = .498, Fisher's Exact Test

16. Secondary Outcome: Incidence of Nocturnal Hypoglycemia (Overall)
Description: Incidence of nocturnal hypoglycemia experienced overall during the study
Time Frame: Baseline to 20 Weeks
Population: As Treated Patients
Measure: Number; unit: Participants
Arm/Group | Exenatide + Placebo | Exenatide + Sitagliptin
Number analyzed (Participants) | 127 | 128
Participants | 0 | 3
Statistical Analysis 1: Comparison: Exenatide + Placebo vs Exenatide + Sitagliptin; Test type: Superiority or Other; p = .247, Fisher's Exact Test

17. Secondary Outcome: Incidence of Confirmed Hypoglycemia(Overall)
Description: Incidence of confirmed hypoglycemia experienced overall during the study
Time Frame: Baseline to 20 Weeks
Population: As Treated Patients; Hypoglycemia defined as: patient experiencing a sign or symptom associated with hypoglycemia that is either self-treated or resolves on its own; has a concurrent fingerstick blood glucose <3.0 mmol/L (54 mg/dL).
Measure: Number; unit: Participants
Arm/Group | Exenatide + Placebo | Exenatide + Sitagliptin
Number analyzed (Participants) | 127 | 128
Participants | 1 | 2
Statistical Analysis 1: Comparison: Exenatide + Placebo vs Exenatide + Sitagliptin; Test type: Superiority or Other; p = 1.00, Fisher's Exact Test

ADVERSE EVENTS:
Arm/Group | Exenatide + Placebo | Exenatide + Sitagliptin
Serious Adverse Events (participants affected / at risk) | 4/127 | 6/128
Other Adverse Events (participants affected / at risk) | 36/127 | 28/128
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Exenatide + Placebo (N=127) | Exenatide + Sitagliptin (N=128)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 1
Lumbar hernia (Gastrointestinal disorders) | 1 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0
Angina unstable (Cardiac disorders) | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Coronary artery disease (Cardiac disorders) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Presyncope (Nervous system disorders) | 0 | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1
Urosepsis (Infections and infestations) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Exenatide + Placebo (N=127) | Exenatide + Sitagliptin (N=128)
Nausea (Gastrointestinal disorders) | 20 | 13
Vomiting (Gastrointestinal disorders) | 13 | 4
Nasopharyngitis (Infections and infestations) | 11 | 10
Headache (Nervous system disorders) | 6 | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days